CLINICAL TRIAL: NCT02159521
Title: ACCElerated ThrombolySiS for Post-Thrombotic Syndrome Using the EKOS System
Brief Title: Treatment of Chronic Deep Vein Thrombosis (DVT) and Post-Thrombotic Syndrome (PTS) With the EkoSonic® Endovascular System
Acronym: ACCESS PTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKOS-11
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Deep Vein Thrombosis; Post-thrombotic Syndrome
Keywords: deep vein thrombosis; post-thrombotic syndrome; chronic deep vein thrombosis
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EkoSonic® Endovascular System (Experimental): Thrombolytic infusion (Alteplase), at an infusion rate of 0.5-1.0 milligrams/hour (mg/hr) will be delivered to the participants with chronic lower extremity venous obstruction after DVT and PTS through the EkoSonic® Endovascular System for at least 12 hours and overnight as needed up to a maximum of 48 hrs. The alteplase dose could be adjusted per investigator discretion, but not to be exceeded 1 mg/hr or a total dose of 48 mg.
  Interventions: Device: EkoSonic® Endovascular System; Biological: Alteplase

INTERVENTIONS:
Device: EkoSonic® Endovascular System
Biological: Alteplase — Recombinant tissue plasminogen activator

SUMMARY:
To evaluate the efficacy of ultrasound accelerated thrombolysis using the EkoSonic® Endovascular System with standard infusion of thrombolytic drug for post-thrombotic syndrome from chronic venous occlusion.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety and efficacy of ultrasound accelerated thrombolysis using the EkoSonic® Endovascular System with standard infusion of a thrombolytic drug for PTS and chronic DVT. Clinical effectiveness will be evaluated using a standard measure of severity of post-thrombotic syndrome over a year.

ELIGIBILITY:
Key Inclusion criteria:

1. Male or female greater than or equal to (≥) 18 years of age and less than or equal to (≤) 75 years of age.
2. Proximal DVT (iliac vein, common femoral vein, deep femoral vein, and femoral vein) that was objectively diagnosed with duplex imaging and/or venography ≥ 6 months prior to study screening.
3. Persistent chronic DVT causing restrictive flow, as confirmed by imaging, within 60 days prior to the study procedure.
4. Villalta score ≥8 for the affected limb within 30 days prior to the study procedure.
5. Failed a minimum of 3 consecutive months of conservative treatment (therapeutic anticoagulation and compression stockings) according to the completed Adherence to Conservative Treatment Form.

Key Exclusion Criteria:

1. Treated with mechanical thrombectomy within 2 weeks of the study thrombolysis procedure.
2. Treated with thrombolysis drugs within 48 hours of the study thrombolytic procedure.
3. Life expectancy less than (<) 1 year.
4. Body Mass Index (BMI) greater than (>) 40 kilograms/square meter (kg/m^2) or per Investigator's discretion participant is able tolerate the procedure and be compliant with post-procedure increased physical activity.
5. No flow in popliteal vein on duplex imaging
6. Isolated iliac vein only thrombus.
7. Thrombus extending ≥ 3 centimeters (cm) into the inferior vena cava (IVC). If central venous occlusion, consider computed tomography (CT) or magnetic resonance venography (MRV). For participants with bilateral DVT, it is recommended that central imaging be performed prior to treatment to evaluate the status of the IVC.
8. Active bleeding, recent (<3 months) gastrointestinal (GI) bleeding, active peptic ulcer, severe liver dysfunction, and bleeding diathesis.
9. Recent (<3 months) internal eye surgery or hemorrhagic retinopathy; recent (<10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation (CPR), obstetrical delivery, or other invasive procedure.
10. History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, or aneurysm.
11. Active cancer (metastatic, progressive, or treated within the last 6 months). Participants with non-melanoma primary skin cancers are eligible to participate in the study.
12. Hemoglobin <9.0 milligrams/deciliter (mg/dL) within 24 hours prior to the procedure
13. International normalized ratio (INR) ≥1.5 nanograms/deciliter (ng/dL) within 24 hours prior to the procedure.
14. Platelet count <100,000 cells/cubic millimeter (cells/mm^3) or >700,000 cells/mm^3 within 24 hours prior to the procedure.
15. Creatinine outside the normal range for the treating institution and considered clinically significant by the Investigator.
16. Uncontrolled hypertension, defined as systolic >175 millimeters of mercury (mmHg) and a diastolic >110 mmHg.
17. Use of clopidogrel, ticlopidine, or other thienopyridine antiplatelet drug within 7 days of the study procedure.
18. In the judgment of the clinician, the participant is at high risk for catastrophic bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Garcia, MD, Principal Investigator — Wilmington DE
Locations (22):
- United States (22):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Vascular Breakthroughs, Darien, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - CHI Health St. Elizabeth, Lincoln, Nebraska
  - Holy Name Medical Center, Teaneck, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Aultman Hospital, Canton, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - DFW Vascular Group/ Methodist Dallas Medical Ctr, Dallas, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia MJ, Sterling KM, Kahn SR, Comerota AJ, Jaff MR, Ouriel K, Weinberg I; ACCESS PTS Investigators. Ultrasound-Accelerated Thrombolysis and Venoplasty for the Treatment of the Postthrombotic Syndrome: Results of the ACCESS PTS Study. J Am Heart Assoc. 2020 Feb 4;9(3):e013398. doi: 10.1161/JAHA.119.013398. Epub 2020 Jan 25. PMID 31983322
- See also: study website — http://www.chronicdvtstudy.com
- See also: EKOS company website — http://www.ekoscorp.com

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Limbs
Groups:
- EkoSonic® Endovascular System: Thrombolytic infusion (Alteplase), at an infusion rate of 0.5-1.0 milligrams/hour (mg/hr) was delivered to the participants with chronic lower extremity venous obstruction after deep vein thrombosis (DVT) and post-thrombotic syndrome (PTS), through EkoSonic® Endovascular System for at least 12 hours and overnight as needed up to a maximum of 48 hrs. The alteplase dose could have been adjusted per investigator discretion, but was not exceeded 1 mg/hr or a total dose of 48 mg.
Period: Overall Study
Arm/Group | EkoSonic® Endovascular System
Started | 81; 85 Limbs (4 participants had both limbs treated.)
Received EkoSonic® Treatment | 78; 82 Limbs
Completed | 63; 67 Limbs
Not Completed | 18; 18 Limbs
Not completed — Enrolled but not treated | 3
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 6
Not completed — Death | 1
Not completed — Other than specified | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Groups:
- EkoSonic® Endovascular System: Thrombolytic infusion (Alteplase), at an infusion rate of 0.5-1.0 mg/hr was delivered to the participants with chronic lower extremity venous obstruction after DVT and PTS, through EkoSonic® Endovascular System for at least 12 hours and overnight as needed up to a maximum of 48 hrs. The alteplase dose could have been adjusted per investigator discretion, but was not exceeded 1 mg/hr or a total dose of 48 mg.
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, not of Hispanic origin | 58
  African American, not of Hispanic origin | 12
  Hispanic or Latino | 5
  Asian or Pacific Islander | 1
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Villalta Score at Day 30 Post-EkoSonic® Study Treatment Procedure
Description: Clinical efficacy was evaluated using the Villalta score at Baseline compared to 30 days Post-EkoSonic® study treatment procedure. Villalta scale (post thrombotic syndrome score) is used for the assessment of symptoms and clinical signs. Participants rated the following symptoms for each leg: pain, cramps, heaviness, pruritus, and paresthesia on a scale ranging from 0 (not present/minimal) to 3 (severe). The study coordinator or nurse rated the following clinical signs in participants for each leg: pre-tibial edema, induration of the skin, hyperpigmentation, new venous extasia, redness during calf compression, and pain during calf compression on a scale ranging from 0 (not present/minimal) to 3 (severe). Total score ranged from 0 to 33. Higher scores represent more severe disease.
Time Frame: Baseline (within 30 days of treatment), Day 30
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated. Here, 'Number analyzed' signifies number of limbs analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Number analyzed (Limbs) | 82
units on a scale
  Baseline | 15.5 (5.17)
  Change at Day 30: number analyzed (Limbs) | 79
  Change at Day 30 | -5.9 (5.75)

2. Primary Outcome: Percentage of Segments of Limbs That Achieved at Least 4-Point Reduction From Baseline in Villalta Score at Day 30
Description: Clinical efficacy was evaluated using the Villalta score at Baseline compared to 30 days Post-EkoSonic® study treatment procedure. Limbs with revascularization procedures were considered non-responders. Villalta scale (post thrombotic syndrome score) is used for the assessment of symptoms and clinical signs. Participants rated the following symptoms for each leg: pain, cramps, heaviness, pruritus, and paresthesia on a scale ranging from 0 (not present/minimal) to 3 (severe). The study coordinator or nurse rated the following clinical signs in participants for each leg: pre-tibial edema, induration of the skin, hyperpigmentation, new venous extasia, redness during calf compression, and pain during calf compression on a scale ranging from 0 (not present/minimal) to 3 (severe). Total score ranged from 0 to 33. Higher scores represent more severe disease.
Time Frame: Baseline (within 30 days of treatment), Day 30
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of segments
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 75
Number analyzed (Limbs) | 79
percentage of segments | 64 [54 to 74]

3. Primary Outcome: Change From Baseline in Blood Flow (Calculated by Time to Washout in the Affected Segment) at Post-Adjunctive Therapy
Description: Change in blood flow was calculated by time to washout in the affected segments in the participants. Time to femoral vein (FV) washout and external iliac vein (EIV) washout was reported.
Time Frame: Baseline (Within 30 days of treatment), Day 0
Population: ITT population included all enrolled participants for whom EkoSonic® treatment was initiated. Here, 'Overall number of participants analyzed'/'Overall Number of Units Analyzed' signifies the number of participants/units evaluable for this outcome measure and 'Number analyzed' signifies number of limbs/participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 49
Number analyzed (Limbs) | 50
seconds
  FV washout: Baseline | 4.39 (2.55)
  FV washout: Change at Day 0: number analyzed (Participants) | 31
  FV washout: Change at Day 0: number analyzed (Limbs) | 31
  FV washout: Change at Day 0 | -2.17 (2.24)
  EIV washout: Baseline: number analyzed (Participants) | 45
  EIV washout: Baseline: number analyzed (Limbs) | 45
  EIV washout: Baseline | 3.28 (2.73)
  EIV washout: Change at Day 0: number analyzed (Participants) | 24
  EIV washout: Change at Day 0: number analyzed (Limbs) | 24
  EIV washout: Change at Day 0 | -0.96 (2.99)

4. Primary Outcome: Number of Participants With Major Bleeding
Description: Major bleeding was defined as: Fatal bleeding; and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome; and/or bleeding causing a fall in hemoglobin of ≥2.0 grams/deciliter (g/dL), or leading to transfusion of ≥2 units of whole blood or red blood cells. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From start of study drug infusion up to 72 hours
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Participants | 1

5. Secondary Outcome: Change From Baseline in Ouriel Score (Venous Volumetric Index [VVI]) at Post-Adjunctive Therapy
Description: The Ouriel score was designed to provide a more accurate quantitative estimate of the thrombus mass by calculating a volumetric index for all the venous segments. 10 venous segments were considered. Included segments were the inferior vena cava, common iliac veins, external iliac veins, internal iliac veins, common femoral veins, superficial and deep femoral veins, and popliteal veins and segments of the anterior tibial veins, posterior tibial veins, and peroneal veins. A normalized volumetric score was calculated for each segment by combining measurements from computed tomography, ultrasonography, and venography. Partially occluded veins were assigned a score of one-half the score value for the segment. The score varies from 1 for a single calf vein to 26 for the infrarenal inferior vena cava. The maximum score was 63 per limb. Higher score indicated worse disease prognoses.
Time Frame: Baseline (Within 30 days of treatment), Day 0
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 68
Number analyzed (Limbs) | 71
units on a scale
  Baseline | 10.58 (6.25)
  Change at Post-EkoSonic® procedure: number analyzed (Participants) | 54
  Change at Post-EkoSonic® procedure: number analyzed (Limbs) | 56
  Change at Post-EkoSonic® procedure | 6.88 (5.69)

6. Secondary Outcome: Number of Participants With at Least 5-Point Reduction From Baseline in Ouriel Score at Post-Adjunctive Therapy
Description: The Ouriel score was designed to provide a more accurate quantitative estimate of the thrombus mass by calculating a volumetric index for all the venous segments. 14 venous segments were considered. Included segments were the inferior vena cava, common iliac veins, external iliac veins, internal iliac veins, common femoral veins, superficial femoral veins, deep femoral veins, and popliteal veins and segments of the anterior tibial veins, posterior tibial veins, and peroneal veins. A normalized volumetric score was calculated for each segment by combining measurements from computed tomography, ultrasonography, and venography. Partially occluded veins were assigned a score of one-half the score value for the segment. The score varies from 1 for a single calf vein to 26 for the infrarenal inferior vena cava. The maximum score was 63 per limb. Higher score indicated worse disease prognoses.
Time Frame: Baseline (Within 30 days of treatment), Day 0
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated. Here, 'Number analyzed' signifies number of participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 54
Participants | 0

7. Secondary Outcome: Change From Baseline in Villalta Score at Days 90, 180, and 365 Post-EkoSonic® Study Treatment Procedure
Description: Villalta scale (post thrombotic syndrome score) is used for the assessment of symptoms and clinical signs. Participants rated the following symptoms for each leg: pain, cramps, heaviness, pruritus, and paresthesia on a scale ranging from 0 (not present/minimal) to 3 (severe). The study coordinator or nurse rated the following clinical signs in participants for each leg: pre-tibial edema, induration of the skin, hyperpigmentation, new venous extasia, redness during calf compression, and pain during calf compression on a scale ranging from 0 (not present/minimal) to 3 (severe). Total score ranged from 0 to 33. Higher scores represent more severe disease.
Time Frame: Baseline (within 30 days of treatment), Days 90, 180, and 365
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated. Here, 'Number analyzed' signifies number of limbs and the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Number analyzed (Limbs) | 82
units on a scale
  Baseline | 15.5 (5.17)
  Change at Day 90: number analyzed (Participants) | 70
  Change at Day 90: number analyzed (Limbs) | 74
  Change at Day 90 | -6.9 (6.48)
  Change at Day 180: number analyzed (Participants) | 66
  Change at Day 180: number analyzed (Limbs) | 69
  Change at Day 180 | -7.8 (6.09)
  Change at Day 365: number analyzed (Participants) | 62
  Change at Day 365: number analyzed (Limbs) | 66
  Change at Day 365 | -8.2 (6.43)

8. Secondary Outcome: Percentage of Segments of Limbs That Achieved at Least 4-Point Reduction From Baseline in Villalta Score at Days 90, 180, and 365
Description: Limbs with revascularization procedures were considered non-responders. Villalta scale (post thrombotic syndrome score) is used for the assessment of symptoms and clinical signs. Participants rated the following symptoms for each leg: pain, cramps, heaviness, pruritus, and paresthesia on a scale ranging from 0 (not present/minimal) to 3 (severe). The study coordinator or nurse rated the following clinical signs in participants for each leg: pre-tibial edema, induration of the skin, hyperpigmentation, new venous extasia, redness during calf compression, and pain during calf compression on a scale ranging from 0 (not present/minimal) to 3 (severe). Total score ranged from 0 to 33. Higher scores represent more severe disease.
Time Frame: Baseline (within 30 days of treatment), Days 90, 180, and 365
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of segments
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 70
Number analyzed (Limbs) | 74
percentage of segments
  Day 90 | 66 [55 to 76]
  Day 180: number analyzed (Participants) | 66
  Day 180: number analyzed (Limbs) | 69
  Day 180 | 74 [62 to 84]
  Day 365: number analyzed (Participants) | 62
  Day 365: number analyzed (Limbs) | 66
  Day 365 | 74 [62 to 84]

9. Secondary Outcome: Percentage of Treated Veins Segments of Limbs With Absence of Re-Occlusion, as Documented by Duplex Imaging
Description: Absence of re-occlusion in following treated veins has been reported: common femoral vein (CFV), common iliac vein (CIV), distal femoral vein (FV), external iliac vein (EIV), popliteal vein, and proximal femoral vein (FV).
Time Frame: Day 365
Population: as for outcome 3
Measure: Number; unit: percentage of segments
Units Other Than Participants: Vein segments
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 51
Number analyzed (Vein segments) | 63
percentage of segments
  CFV: number analyzed (Participants) | 43
  CFV: number analyzed (Vein segments) | 44
  CFV | 100
  CIV: number analyzed (Participants) | 14
  CIV: number analyzed (Vein segments) | 15
  CIV | 100
  Distal FV: number analyzed (Vein segments) | 55
  Distal FV | 100
  EIV: number analyzed (Participants) | 20
  EIV: number analyzed (Vein segments) | 21
  EIV | 100
  Popliteal Vein: number analyzed (Participants) | 44
  Popliteal Vein: number analyzed (Vein segments) | 46
  Popliteal Vein | 97.9
  Proximal FV: number analyzed (Participants) | 47
  Proximal FV: number analyzed (Vein segments) | 51
  Proximal FV | 100

10. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Sub-Scale Score and Physical Component Score (PCS) at Days, 30, 90, 180, and 365
Description: SF- 36 investigates the standard of quality of life through a general health assessment. It is a 36-item questionnaire measuring 8 domains (physical functioning [PF], role physical [RP], bodily pain [BP], general health [GH], vitality [VT], social functioning [SF], role emotional [RE], and mental health [MH]). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. The PCS score summarizes the subscales physical functioning, role-physical, bodily pain, and general health. Total score range for PCS was 0 (lowest level of physical functioning) to 100 (highest level of physical functioning).
Time Frame: Baseline (within 30 days of treatment), Days 30, 90, 180, and 365
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Number analyzed (Limbs) | 82
units on a scale
  PF Score: Baseline | 48.4 (27.75)
  PF Score: Change at Day 30: number analyzed (Participants) | 75
  PF Score: Change at Day 30: number analyzed (Limbs) | 79
  PF Score: Change at Day 30 | 9.5 (21.72)
  PF Score: Change at Day 90: number analyzed (Participants) | 69
  PF Score: Change at Day 90: number analyzed (Limbs) | 73
  PF Score: Change at Day 90 | 14.0 (22.87)
  PF Score: Change at Day 180: number analyzed (Participants) | 68
  PF Score: Change at Day 180: number analyzed (Limbs) | 71
  PF Score: Change at Day 180 | 15.1 (24.75)
  PF Score: Change at Day 365: number analyzed (Participants) | 61
  PF Score: Change at Day 365: number analyzed (Limbs) | 65
  PF Score: Change at Day 365 | 13.9 (23.40)
  RP Score: Baseline | 47.2 (26.84)
  RP Score: Change at Day 30: number analyzed (Participants) | 75
  RP Score: Change at Day 30: number analyzed (Limbs) | 79
  RP Score: Change at Day 30 | 7.1 (27.86)
  RP Score: Change at Day 90: number analyzed (Participants) | 69
  RP Score: Change at Day 90: number analyzed (Limbs) | 73
  RP Score: Change at Day 90 | 17.6 (23.65)
  RP Score: Change at Day 180: number analyzed (Participants) | 68
  RP Score: Change at Day 180: number analyzed (Limbs) | 71
  RP Score: Change at Day 180 | 19.5 (27.47)
  RP Score: Change at Day 365: number analyzed (Participants) | 61
  RP Score: Change at Day 365: number analyzed (Limbs) | 65
  RP Score: Change at Day 365 | 17.6 (28.42)
  BP Score: Baseline | 46.2 (25.44)
  BP Score: Change at Day 30: number analyzed (Participants) | 75
  BP Score: Change at Day 30: number analyzed (Limbs) | 79
  BP Score: Change at Day 30 | 6.9 (27.92)
  BP Score: Change at Day 90: number analyzed (Participants) | 69
  BP Score: Change at Day 90: number analyzed (Limbs) | 73
  BP Score: Change at Day 90 | 14.4 (28.04)
  BP Score: Change at Day 180: number analyzed (Participants) | 68
  BP Score: Change at Day 180: number analyzed (Limbs) | 71
  BP Score: Change at Day 180 | 15.2 (29.26)
  BP Score: Change at Day 365: number analyzed (Participants) | 61
  BP Score: Change at Day 365: number analyzed (Limbs) | 65
  BP Score: Change at Day 365 | 16.0 (28.92)
  GH Score: Baseline | 58.6 (22.38)
  GH Score: Change at Day 30: number analyzed (Participants) | 75
  GH Score: Change at Day 30: number analyzed (Limbs) | 79
  GH Score: Change at Day 30 | 1.1 (17.17)
  GH Score: Change at Day 90: number analyzed (Participants) | 69
  GH Score: Change at Day 90: number analyzed (Limbs) | 73
  GH Score: Change at Day 90 | 3.4 (16.10)
  GH Score: Change at Day 180: number analyzed (Participants) | 68
  GH Score: Change at Day 180: number analyzed (Limbs) | 71
  GH Score: Change at Day 180 | 0.8 (15.56)
  GH Score: Change at Day 365: number analyzed (Participants) | 61
  GH Score: Change at Day 365: number analyzed (Limbs) | 65
  GH Score: Change at Day 365 | 0.1 (18.10)
  VT Score: Baseline | 50.5 (23.18)
  VT Score: Change at Day 30: number analyzed (Participants) | 75
  VT Score: Change at Day 30: number analyzed (Limbs) | 79
  VT Score: Change at Day 30 | 2.8 (24.53)
  VT Score: Change at Day 90: number analyzed (Participants) | 69
  VT Score: Change at Day 90: number analyzed (Limbs) | 73
  VT Score: Change at Day 90 | 8.9 (19.35)
  VT Score: Change at Day 180: number analyzed (Participants) | 68
  VT Score: Change at Day 180: number analyzed (Limbs) | 71
  VT Score: Change at Day 180 | 6.6 (21.83)
  VT Score: Change at Day 365: number analyzed (Participants) | 61
  VT Score: Change at Day 365: number analyzed (Limbs) | 65
  VT Score: Change at Day 365 | 5.7 (20.81)
  SF Score: Baseline | 65.4 (31.81)
  SF Score: Change at Day 30: number analyzed (Participants) | 75
  SF Score: Change at Day 30: number analyzed (Limbs) | 79
  SF Score: Change at Day 30 | 2.7 (30.14)
  SF Score: Change at Day 90: number analyzed (Participants) | 69
  SF Score: Change at Day 90: number analyzed (Limbs) | 73
  SF Score: Change at Day 90 | 11.3 (24.40)
  SF Score: Change at Day 180: number analyzed (Participants) | 68
  SF Score: Change at Day 180: number analyzed (Limbs) | 71
  SF Score: Change at Day 180 | 9.9 (27.05)
  SF Score: Change at Day 365: number analyzed (Participants) | 61
  SF Score: Change at Day 365: number analyzed (Limbs) | 65
  SF Score: Change at Day 365 | 9.0 (24.06)
  RE Score: Baseline | 70.8 (30.77)
  RE Score: Change at Day 30: number analyzed (Participants) | 75
  RE Score: Change at Day 30: number analyzed (Limbs) | 79
  RE Score: Change at Day 30 | 3.8 (33.83)
  RE Score: Change at Day 90: number analyzed (Participants) | 69
  RE Score: Change at Day 90: number analyzed (Limbs) | 73
  RE Score: Change at Day 90 | 10.6 (28.30)
  RE Score: Change at Day 180: number analyzed (Participants) | 68
  RE Score: Change at Day 180: number analyzed (Limbs) | 71
  RE Score: Change at Day 180 | 9.9 (27.90)
  RE Score: Change at Day 365: number analyzed (Participants) | 61
  RE Score: Change at Day 365: number analyzed (Limbs) | 65
  RE Score: Change at Day 365 | 3.9 (31.11)
  MH Score: Baseline | 67.5 (21.58)
  MH Score: Change at Day 30: number analyzed (Participants) | 75
  MH Score: Change at Day 30: number analyzed (Limbs) | 79
  MH Score: Change at Day 30 | 3.4 (17.70)
  MH Score: Change at Day 90: number analyzed (Participants) | 69
  MH Score: Change at Day 90: number analyzed (Limbs) | 73
  MH Score: Change at Day 90 | 7.7 (16.54)
  MH Score: Change at Day 180: number analyzed (Participants) | 68
  MH Score: Change at Day 180: number analyzed (Limbs) | 71
  MH Score: Change at Day 180 | 7.2 (19.12)
  MH Score: Change at Day 365: number analyzed (Participants) | 61
  MH Score: Change at Day 365: number analyzed (Limbs) | 65
  MH Score: Change at Day 365 | 4.5 (20.77)
  PCS Score: Baseline | 38.6 (9.47)
  PCS Score: Change at Day 30: number analyzed (Participants) | 75
  PCS Score: Change at Day 30: number analyzed (Limbs) | 79
  PCS Score: Change at Day 30 | 2.8 (7.62)
  PCS Score: Change at Day 90: number analyzed (Participants) | 69
  PCS Score: Change at Day 90: number analyzed (Limbs) | 73
  PCS Score: Change at Day 90 | 5.1 (8.52)
  PCS Score: Change at Day 180: number analyzed (Participants) | 68
  PCS Score: Change at Day 180: number analyzed (Limbs) | 71
  PCS Score: Change at Day 180 | 5.4 (9.24)
  PCS Score: Change at Day 365: number analyzed (Participants) | 61
  PCS Score: Change at Day 365: number analyzed (Limbs) | 65
  PCS Score: Change at Day 365 | 5.8 (8.80)

11. Secondary Outcome: Number of Treated Limbs With Shift From Baseline in Clinical Stages (Symptomatic and Asymptomatic) of Clinical, Etiologic, Anatomic, Pathophysiological (CEAP) Classification at Days 30, 90, 180, and 365
Description: Status of clinical signs and symptoms of lower limb venous disease was measured by CEAP classification. The CEAP clinical Categories were as follows: C0- no visible or palpable signs of venous disease, C1- telangiectasies or reticular veins, C2- varicose veins, C3- edema, C4a- pigmentation and eczema, C4b- lipodermatosclerosis and atrophie blanche, C5- healed venous ulcer, and C6- active venous ulcer. C0 was of the least clinical concern and C6 was the worst stage. Each clinical class was further characterized by the (clinical stages) presence or absence of symptoms (ache, pain, tightness, skin irritation, heaviness, muscle cramps, as well as other complaints attributable to venous dysfunction): asymptomatic and symptomatic.
Time Frame: Baseline (within 30 days of treatment), Days 30, 90, 180, and 365
Population: as for outcome 3
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 75
Number analyzed (Limbs) | 79
Limbs
  Baseline to Day 30: Symptomatic - Symptomatic | 67
  Baseline to Day 30: Symptomatic - Asymptomatic | 12
  Baseline to Day 90: number analyzed (Participants) | 71
  Baseline to Day 90: number analyzed (Limbs) | 75
  Baseline to Day 90: Symptomatic - Symptomatic | 56
  Baseline to Day 90: Symptomatic - Asymptomatic | 19
  Baseline to Day 180: number analyzed (Participants) | 67
  Baseline to Day 180: number analyzed (Limbs) | 70
  Baseline to Day 180: Symptomatic - Symptomatic | 45
  Baseline to Day 180: Symptomatic - Asymptomatic | 25
  Baseline to Day 365: number analyzed (Participants) | 61
  Baseline to Day 365: number analyzed (Limbs) | 65
  Baseline to Day 365: Symptomatic - Symptomatic | 40
  Baseline to Day 365: Symptomatic - Asymptomatic | 25

12. Secondary Outcome: Change From Baseline in Venous Insufficiency Epidemiological and Economic Study Quality of Life (VEINES-QOL) Score At Days 30, 90, 180, and 360
Description: The VEINES-QOL/Sym is a participant-based questionnaire designed for self-completion and measures deep vein thrombosis (DVT) impact on symptoms and quality of life from the participants' perspective. It contains 26 items covering participant DVT: symptoms, limitations in daily activities, and psychological impact. A separate summary score VEINES-QOL ranges from 0 (worst quality of life) to 100 (best quality of life). Higher scores indicated a better quality of life.
Time Frame: Baseline (within 30 days of treatment), Days 30, 90, 180, and 365
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 63
units on a scale
  Baseline | 61.1 (19.63)
  Change at Day 30: number analyzed (Participants) | 62
  Change at Day 30 | 10.3 (15.86)
  Change at Day 90: number analyzed (Participants) | 58
  Change at Day 90 | 16.3 (17.96)
  Change at Day 180: number analyzed (Participants) | 55
  Change at Day 180 | 18.9 (16.23)
  Change at Day 365: number analyzed (Participants) | 53
  Change at Day 365 | 18.7 (16.27)

13. Secondary Outcome: Change From Baseline in Venous Clinical Severity Score (VCSS) in Study Leg at Days 30, 90, 180, and 365
Description: The VCSS system includes 10 clinical descriptions (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, duration of active ulceration, size of active ulceration, and level of compliance with medical compression therapy), scored from 0 to 3 (total possible score, 30) with 0 = absent, 1 = mild, 2 = moderate and 3 = severe. Total VCSS was the sum of all VCSS assessment scores from categories for a given time point. Total score ranged from 0 (absent) to 30 (severe). Lower values represent a better outcome, that is, a level of pain less than that experienced at baseline.
Time Frame: Baseline (within 30 days of treatment), Days 30, 90, 180, and 365
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Limbs
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Number analyzed (Limbs) | 82
units on a scale
  Baseline | 12.0 (5.33)
  Change at Day 30: number analyzed (Participants) | 75
  Change at Day 30: number analyzed (Limbs) | 79
  Change at Day 30 | -3.8 (4.33)
  Change at Day 90: number analyzed (Participants) | 69
  Change at Day 90: number analyzed (Limbs) | 73
  Change at Day 90 | -4.5 (4.97)
  Change at Day 180: number analyzed (Participants) | 67
  Change at Day 180: number analyzed (Limbs) | 70
  Change at Day 180 | -5.2 (4.68)
  Change at Day 365: number analyzed (Participants) | 60
  Change at Day 365: number analyzed (Limbs) | 64
  Change at Day 365 | -5.7 (4.38)

14. Secondary Outcome: Number of Participants With PTS-induced Admission to an Emergency Room or Unplanned Visits to a Physician's Office or Hospitalization
Description: Number of participants with PTS-induced admission to an emergency room or unplanned visits to a physician's office or hospitalization, are reported. A participant can have more than one PTS-induced health issue.
Time Frame: From the time of the EkoSonic® procedure (Day 0) up to 365 days
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Participants
  Total | 24
  Emergency Room | 13
  Unplanned Physician Office Visit | 18
  Hospitalization | 8

15. Secondary Outcome: Time From Starting Initial Thrombolytic Infusion to Discharge From the Hospital
Description: This Outcome Measure was to measure the time that the participant's initial thrombolytic infusion started to the time the participant was discharged from the hospital.
Time Frame: From the time of the EkoSonic® procedure (Day 0) up to 365 days
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Measure: Median (Full Range); unit: days
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
days | 2 [1 to 38]

16. Secondary Outcome: Number of Participants Who Had Symptomatic PE During Hospitalization for Study Procedure
Description: Symptomatic PE was diagnosed using computed tomography pulmonary angiogram (CTPA), single positron emission computed tomography (SPECT), and ventilation-perfusion (VQ).
Time Frame: From starting the initial thrombolytic infusion (Day 0) through discharge from hospital (up to Day 38)
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Participants | 0

17. Secondary Outcome: Number of Participants Who Died Due to Any Cause
Description: Number of participants who died due to any cause for up to 365 days following the conclusion of the study procedure, were reported.
Time Frame: Baseline (within 30 days of treatment) up to Day 365
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Participants | 1

18. Secondary Outcome: Number of Participants Who Had Adverse Events (AEs), Related (to the Study Procedure/Device/Medications) AEs, and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A summary of non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (within 30 days of treatment) up to Day 30
Population: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | EkoSonic® Endovascular System
Number analyzed (Participants) | 78
Participants
  Any AEs | 34
  Related to Thrombolytic/Angiographic Procedure | 15
  Related to EKOS system | 3
  Related to Thrombolytic Drug | 8
  Related to Anticoagulant Drug | 15
  Related to Post-procedure Adjunctive Treatment | 3
  SAEs | 12

ADVERSE EVENTS:
Time Frame: Baseline (within 30 days of treatment) up to Day 365
Description: ITT population included all enrolled participants for whom the EkoSonic® treatment was initiated.
Arm/Group | EkoSonic® Endovascular System
All-Cause Mortality (participants affected / at risk) | 1/78
Serious Adverse Events (participants affected / at risk) | 16/78
Other Adverse Events (participants affected / at risk) | 33/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EkoSonic® Endovascular System (N=78)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Oxygen saturation decreased (Investigations) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 8
Epistaxis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Venous occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EkoSonic® Endovascular System (N=78)
Haematoma (Vascular disorders) | 2
Sinusitis (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 6
Procedural haemorrhage (Injury, poisoning and procedural complications) | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Hypertension (Vascular disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Bradycardia (Cardiac disorders) | 2
Pelvic venous thrombosis (Vascular disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Anxiety (Psychiatric disorders) | 2
Epistaxis (Vascular disorders) | 1
Injection site haemorrhage (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Haemorrhage (Vascular disorders) | 1
Migraine (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Blood fibrinogen decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02159521/Prot_001.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02159521/SAP_000.pdf